CLINICAL TRIAL: NCT05850650
Title: The Effect of Collagen Sponge Placed in the Socket After Surgical Extraction of Mandibular Third Molars on the Incidence of Alveolar Osteitis. A Randomized Controlled Trial
Brief Title: The Effect of Post-extraction Collagen Sponge Application on Alveolar Osteitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Nedal Abu-Mostafa, Assistant Professor in Oral and Maxillofacial Surgery, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REU
Record Dates: First submitted 2023-03-19; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Alveolar Osteitis
Keywords: alveolar osteitis; Collagen sponge; Impacted lower third molar
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: The patients will have surgical extraction of impacted 3rd molars for both sides with a gap of 3 weeks. The study side will receive a collage sponge after extraction followed by sutures. The controlled side will have sutures without a collagen sponge.
Who Masked: Participant
Masking Description: The participants (patients) will not be informed about which side will recieve the collagen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controlled (Active Comparator): The extraction socket will not receive a collagen sponge
  Interventions: Other: No collagen sponge application after surgical extraction of impacted 3rd molar
- Collagen (Experimental): The extraction socket will receive a collagen sponge
  Interventions: Other: Application of a collagen sponge after surgical extraction of impacted 3rd molar

INTERVENTIONS:
Other: Application of a collagen sponge after surgical extraction of impacted 3rd molar — Application of a collagen sponge after surgical extraction of impacted 3rd molar
  Arms: Collagen
Other: No collagen sponge application after surgical extraction of impacted 3rd molar — No collagen sponge application after surgical extraction of impacted 3rd molar
  Arms: Controlled

SUMMARY:
The goal of this randomized controlled trial is to compare pain, mouth opening, and alveolar osteitis following surgical extraction of bilateral symmetrical impacted lower third molars using two types of wound closures. Collagen plugs will be applied in the sockets of the study side followed by suture, while the controlled side will be sutured without a collagen plug. The study will include 40 patients aged between 18- 40 years old, medically fit (ASA1), who have bilateral symmetrical impacted lower third molars and visit the oral surgery clinics of King Saud Medical City for extraction. The main question is" Does intra-alveolar collagen application after surgical extraction of impacted lower third molars reduce the incidence of alveolar osteitis?

ELIGIBILITY:
Inclusion Criteria:

Forty patients aged between 18- 40 years old, ASA1, who have bilateral symmetrical impacted lower third molars and visit the oral surgery clinics of King Saud Medical City for extraction.

Exclusion Criteria:

Uncontrolled systemic diseases, diabetes, bone diseases, smokers, epinephrine contraindications, pregnant women, breastfeeding women, and those who were using oral contraceptives.

Other exclusion criteria are the presence of acute infection and facial swelling, cystic lesions, and TMJ problems. Moreover, any surgical extraction that lasts more than 30 minutes +/- 5 minutes, or has been done without the whole standardized steps will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Pre-extraction Pain score | Pre-extraction
  Pain measurement by VAS (0-10). 0: no pain. 10: worst pain
Pre-extraction Halitosis | Pre-extraction
  Halitosis in reported in the presence of a bad odor that is smelled by the investigator during the patient's speech
Pre-extraction Mouth opening | Pre-extraction
  Maximum Mouth opening is taken by a caliber
Pain score Day3 | 3 days after extraction
  Pain measurement by VAS (0-10). 0: no pain. 10: worst pain
Pain score Day7 | 7 days after extraction
  Pain measurement by VAS (0-10). 0: no pain. 10: worst pain
Mouth opening Day7 | 7 days after extraction
  Maximum Mouth opening is taken by a caliber
Halitosis Day7 | 7 days after extraction
  Halitosis in reported in the presence of a bad odor that is smelled by the investigator during the patient's speech
Alveolar osteitis | After 3 days of extraction
  is diagnosed if the patient complains of pain (more than 5) between day 2 and day 4 with empty sockets and food debris, with or without halitosis

CONTACTS AND LOCATIONS:
Overall Officials: Nedal A Abu-Mostafa, Assistant P, Principal Investigator — nabumostafa@gmail.com
Locations (1):
- RiyadH Colleges of dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
It will be available in the published manuscript